CLINICAL TRIAL: NCT05900206
Title: A Randomized Trial of Trastuzumab Deruxtecan and Biology-Driven Selection of Neoadjuvant Treatment for HER2-positive Breast Cancer: ARIADNE
Brief Title: Trastuzumab Deruxtecan Versus Standard Neoadjuvant Treatment for HER2-positive Breast Cancer
Acronym: ARIADNE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Theodoros Foukakis, Associate Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARIADNE
Record Dates: First submitted 2023-05-21; First posted 2023-06-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: HER2-positive; neoadjuvant treatment; trastuzumab deruxtecan; T-DXd; PAM50; molecular subtype; ribociclib; HER2-enriched; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; Docetaxel; Paclitaxel; Carboplatin; Trastuzumab; pertuzumab; ribociclib; Letrozole; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Parallel, two arms for cycles 1-3. Further treatment (cycles 4-6) decided by molecular intrinsic subtype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- T-DXd (cycles 1-3) (Experimental): Trastuzumab Deruxtecan, administered every three weeks for three courses. Further treatment is decided by the intrinsic molecular (PAM50) subtype of the tumor.
  Interventions: Drug: Trastuzumab deruxtecan
- Standard treatment (TCHP or PCHP; cycles 1-3) (Active Comparator): TCHP (Docetaxel, Carboplatin, Trastuzumab, Pertuzumab) or PCHP (Paclitaxel, Carboplatin, Trastuzumab, Pertuzumab), administered every three weeks for three courses. Further treatment is decided by the intrinsic molecular (PAM50) subtype of the tumor.
  Interventions: Drug: Docetaxel; Drug: Paclitaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab
- ER-positive and Luminal (cycles 4-6) (Other): Ribociclib, letrozole, trastuzumab, pertuzumab
  Interventions: Drug: Ribociclib; Drug: Letrozole
- ER-negative and Luminal, or Basal-like, or Normal-like (cycles 4-6) (Other): Epirubicin and Cyclophosphamide in case of no complete radiologic response after the initial three courses. In case of complete radiologic response, treatment from cycles 1-3 (T-DXd or TCHP/PCHP) will continue instead for three more courses.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide
- HER2-enriched (cycles 4-6) (Other): The same treatment with T-DXd or TCHP/PCHP administered every three weeks for three more courses will continue from cycles 1-3
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Docetaxel; Drug: Paclitaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Experimental drug. Provided in 100mg vials. IV infusion.
  Other Names: T-DXd, Enhertu
  Arms: HER2-enriched (cycles 4-6); T-DXd (cycles 1-3)
Drug: Docetaxel — Active comparator. IV infusion.
  Arms: HER2-enriched (cycles 4-6); Standard treatment (TCHP or PCHP; cycles 1-3)
Drug: Paclitaxel — Active comparator. IV infusion.
  Arms: HER2-enriched (cycles 4-6); Standard treatment (TCHP or PCHP; cycles 1-3)
Drug: Carboplatin — Active comparator. IV infusion.
  Arms: HER2-enriched (cycles 4-6); Standard treatment (TCHP or PCHP; cycles 1-3)
Drug: Trastuzumab — Active comparator. IV infusion.
  Other Names: Herceptin
  Arms: HER2-enriched (cycles 4-6); Standard treatment (TCHP or PCHP; cycles 1-3)
Drug: Pertuzumab — Active comparator. IV infusion.
  Other Names: PErjeta
  Arms: HER2-enriched (cycles 4-6); Standard treatment (TCHP or PCHP; cycles 1-3)
Drug: Ribociclib — Experimental drug. Tablets.
  Other Names: Kisqali
  Arms: ER-positive and Luminal (cycles 4-6)
Drug: Letrozole — Experimental drug. Tablets.
  Arms: ER-positive and Luminal (cycles 4-6)
Drug: Epirubicin — Active comparator. IV infusion.
  Arms: ER-negative and Luminal, or Basal-like, or Normal-like (cycles 4-6)
Drug: Cyclophosphamide — Active comparator. IV infusion.
  Arms: ER-negative and Luminal, or Basal-like, or Normal-like (cycles 4-6)

SUMMARY:
The goal of this clinical trial is to compare trastuzumab deruxtecan (T-DXd) to standard preoperative treatment in patients with non-metastatic HER2-positive breast cancer. The main questions it aims to answer are:

* is T-DXd more effective than standard preoperative treatment?
* are there markers in the tumor or blood of patients with HER2-positive breast cancer that can help us predict response to treatment?

Participants will be divided into two groups, where one group will be treated with three courses of T-DXd and the other group will be treated with three courses standard of care treatment. Thereafter, further treatment will be decided by the tumor's molecular subtype.

ELIGIBILITY:
To be eligible for the study, patients must fulfil all inclusion criteria:

1. Women or men 18 years or older
2. Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations
3. Histologically confirmed breast cancer with an invasive component measuring ≥ 20 mm and/or with morphologically confirmed spread to regional lymph nodes (stage cT2-cT4 with any cN, or cN1-cN3 with any cT).
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at the time of randomization (see Appendix B).
5. Known estrogen-receptor and/or progesterone receptor status, as assessed locally by IHC. The cut-off for positivity for ER/PR for this study is at least 10% of cell nuclei staining for ER or PR, respectively.
6. Known HER2-positive breast cancer defined as an IHC status of 3+. If IHC is 2+, a positive in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing. ISH positivity is defined as a ratio of ≥ 2 for the number of HER2 gene copies to the number of signals for chromosome 17 copies.
7. Left Ventricular Ejection Fraction (LVEF) ≥ 50%
8. Adequate bone-marrow, hepatic and renal function defined as laboratory tests within 7 days prior to enrolment:

   i. Hematology:
   1. Absolute granulocytes > 1.5 x 109/L
   2. Platelets > 100 x 109/L
   3. Hb > 90 gr/L ii. Biochemistry

   <!-- -->

   1. Bilirubin ≤ upper limit of normal (ULN)
   2. Serum creatinine ≤ 1.5 x ULN
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 x ULN
   4. Albumin ≥ 30 gr/L iii. Coagulation:

   <!-- -->

   1. INR/PT ≤ 1.5 x ULN, unless the subject is receiving anticoagulant therapy and INR/PT is within intended therapeutic range
   2. aPTT ≤ 1.5 x ULN, unless the subject is receiving anticoagulant therapy and aPTT is within intended therapeutic range
9. Availability of tumor and blood samples as described in the protocol
10. Negative serum pregnancy test for women of childbearing potential or for patients who have experienced menopause onset <12 months prior to randomization.
11. Patients of childbearing potential must be willing to use one highly effective contraception or two effective forms of nonhormonal contraception. See also 5.6 Precautions.
12. Participants must be able to communicate with the investigator and comply with the requirements of the study procedures

To be eligible for the study, patients must not fulfil any exclusion criteria:

1. Participation in other interventional trials
2. Presence of distant metastases, including node metastases in the contralateral thoracic region or in the mediastinum
3. Other malignancy diagnosed during the past five years, except adequately controlled limited basal cell carcinoma or squamous-cell carcinoma of the skin, in situ melanoma or carcinoma in situ of the cervix.
4. History of invasive breast cancer
5. History of DCIS, except for patients treated exclusively with mastectomy >5 years prior to diagnosis of current breast cancer
6. Active cardiac disease or a history of cardiac dysfunction including any of the following:

   1. History of unstable angina pectoris, myocardial infarction or recent (<6 months) cardiovascular event including stroke and pericarditis
   2. History of documented congestive heart failure (New York Heart Association functional classification II-IV)
   3. Documented cardiomyopathy
   4. QTc > 450 msec as measured by Fridericia's formula, family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes.
   5. Uncontrolled hypertension
   6. Symptomatic or uncontrolled arrhythmia, including atrial fibrillation.
7. Patients with ER-positive BC being treated with drugs recognized as strong inhibitors or inducers of the isoenzyme CYP3A (see table 5) which cannot be discontinued at least 7 days prior to planned treatment with ribociclib.
8. Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointes that cannot be discontinued or replaced by safe alternative medication
9. Pregnant or breastfeeding female patients, or patients who are planning to become pregnant
10. History of (non-infectious) Interstitial Lung Disease (ILD) / pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
11. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.)
12. Any autoimmune, connective tissue or inflammatory disorders (e.g. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for patients who are included in the study.
13. Prior pneumonectomy
14. History of positive testing for HIV or known AIDS
15. Acute or chronic infection with hepatitis B or C virus
16. Any impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
17. Receipt of live, attenuated vaccine within 30 days prior to the first dose of trastuzumab deruxtecan. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of study drug.
18. Any psychological, including substance abuse, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
19. Allergic reactions or hypersensitivity to the study drugs or other monoclonal antibodies
20. Administration of other experimental drugs, either concomitantly or during the past 30 days before treatment initiation.
21. Pre-treatment axillary surgery
22. Recent major surgery (within 4 weeks from start of study treatment) or anticipated need for major surgery during the study.
23. A pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) of HER2-enriched patients | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Locally assessed rate of pCR at the molecularly HER2-enriched population, defined as ypT0/Tis, ypN0, as determined at the surgical specimen by a pathologist blinded to treatment assignment (intention-to-treat analysis)

SECONDARY OUTCOMES:
Pathologic complete response (pCR) of the initially randomized patients | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Locally assessed rate of pCR, defined as ypT0/Tis, ypN0, at the two patient groups of the initial randomization of TCHP versus T-DXd, regardless of administered therapy after cycle 3
Event-free survival | From randomization to event, up to five years
  Event-free survival (EFS), defined as time from randomization to breast cancer relapse, contralateral breast cancer, other malignant neoplasms, or death by any cause, for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd
Biomarkers | From randomization to event, up to five years
  Exploratory analysis of biomarkers of response/resistance to administered neoadjuvant therapy using genomics, transcriptomics and proteomics in both tumor tissue and blood/plasma
Pathologic complete response (pCR) of ER-positive and luminal patients | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Locally assessed rate of pCR at ER-positive and luminal subgroup
Pathologic complete response (pCR) of ER-negative and luminal, basal-like and normal-like patients | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Locally assessed rate of pCR at ER-negative and luminal subgroup, at the basal-like subgroup and the normal-like subgroup
Objective response rate at three cycles | After the completion of three treatment cycles (each cycle is 21 days)
  Rates of radiologic complete response after three courses of either standard therapy or T-DXd
Overall survival | From randomization to event, up to five years
  Overall survival (OS), defined as time from randomization to death by any cause, for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd
Distant relapse-free survival | From randomization to event, up to five years
  Distant relapse-free survival (DRFS), defined as time from randomization to distant metastases or death by any cause, for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd
Objective response rate at six cycles | After the completion of six treatment cycles (each cycle is 21 days)
  Rates of complete radiologic response, for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd
Residual Cancer Burden | Categorical outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Pathologic response according to Residual Cancer Burden Class for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd
Breast conserving surgery | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Rate of breast conserving surgery, for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd
De-escalation of breast surgery | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Rate of de-escalation of breast surgery (conversion from mastectomy to breast conserving surgery or de-escalation of complexity from an oncoplastic breast-conserving procedure to simple wide local excisions) for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd
Sentinel Lymph Node Dissection | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Rate of Sentinel Lymph Node Dissection (SLND), for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd
De-escalation of axillary surgery | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Rate of de-escalation of axillary surgery (conversion from axillary lymph node dissection to either targeted axillary dissection or sentinel lymph node dissection) for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd
Rates of adverse events | During neoadjuvant treatment at the end of each treatment cycle (cycle length 21 days)
  Frequency and grade of adverse events (AE) (according to NCI CTCAE v. 5.0) and rate of discontinuation due to toxicity
Change From Baseline in Global Health Status/Quality of Life Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in all participants | During neoadjuvant treatment (before first treatment and after three cycles, 21-day cycles), at the end of treatment (after six 21-day cycles), one year post-surgery and five years post-surgery
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score will be presented in all participants. A higher score indicates a better level of function.
Change From Baseline in Physical Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in all participants | During neoadjuvant treatment (before first treatment and after three cycles, 21-day cycles), at the end of treatment (after six 21-day cycles), one year post-surgery and five years post-surgery
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the physical functioning score will be presented in all participants. A higher score indicates a better level of function.
Change From Baseline in Emotional Functioning Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in all participants | During neoadjuvant treatment (before first treatment and after three cycles, 21-day cycles), at the end of treatment (after six 21-day cycles), one year post-surgery and five years post-surgery
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 4 questions about their emotional functioning (Items 21-24) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the emotional functioning score will be presented in all participants. A higher score indicates a better level of function.
Axillary surgery | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Rate of Sentinel Lymph Node detection, Targeted Axillary Dissection success and false-negative rates of these procedures in initially node-positive patients for each molecular group, including the comparison of TCHP versus T-DXd in HER2-enriched patients, and at the two patient groups of the initial randomization of TCHP versus T-DXd

OTHER OUTCOMES:
Exploratory biomarkers | Binary outcome which will be assessed at the time of surgery after six cycles of treatment (each cycle is 21 days)
  Exploratory analyses of clinicopathologic characteristics as predictors for response

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Foukakis, MD/PhD, Principal Investigator — Karolinska University Hospital; Alexios Matikas, MD/PhD, Principal Investigator — Karolinska University Hospital
Locations (7):
- Sweden (7):
  - Skåne University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - Sankt Gorans Hospital, Stockholm
  - Stockholm Southern Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Norrlands University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matikas A, Naume B, Wildiers H, Sonke G, Dieci MV, Karakatsanis A, Andersson A, Barnekow E, Kessler LE, Einbeigi Z, Killander F, Linderholm B, Schiza A, Valachis A, Nearchou A, Engebraaten O, Porojnicu A, Soland MH, Mannsaker B, Raj SX, Blix ES, Nordstrand CS, Lambertini M, Vernieri C, Punie K, Sotiriou C, Bergh J, Villacampa G, Zouzos A, Hellstrom M, Hartman J, Foukakis T. Randomised trial of trastuzumab deruxtecan and biology-driven selection of neoadjuvant treatment for HER2-positive breast cancer: a study protocol of ARIADNE. BMJ Open. 2025 Aug 27;15(8):e102626. doi: 10.1136/bmjopen-2025-102626. PMID 40866060